## Statement of Research – Survey

You are invited to take part in a research study, conducted by the Medical University of South Carolina. The purpose of the study is to help us understand the feasibility and impact of the Be Well Care Well program on early care education teachers, including teacher stress, physical activity, teacher-child interactions, and nutrition. You are being asked to participate because you are employed at the center. Your participation is voluntary, and your participation or discontinuance will not impact any element of your job performance/evaluation and will not become a part of your employment record.

If you decide to participate, your individual answers will be kept strictly confidential, but the overall results of the survey will be used to evaluate the impact of the Be Well Care Well program. There is no penalty if you do not participate. You can skip questions you don't want to answer or end the survey at any time. The survey should take up to 30 minutes to complete and your responses are confidential. There is a risk of loss of confidentiality by completing the survey. You are not expected to personally benefit from completing the survey, but information will be used to improve overall teacher well-being.

You will receive \$25 for completing the pre survey and \$50 for the post survey. Completing the survey implies consent to participate in the research.

If you have any questions about the survey or about research subjects' rights, please contact the Principal Investigator, Dr. Angela Moreland at <a href="mailto:moreland@musc.edu">moreland@musc.edu</a>.

IRB Number: Pro00105341 Date Approved 5/18/2022

